CLINICAL TRIAL: NCT05493150
Title: Antalgic Effects of Well-being Treatments in Cancer Care; Foot Reflexology, Socio-aesthetics, Sophrology, Singing
Brief Title: Antalgic Effects of Well-being Treatments in Cancer Care
Acronym: Well Being
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-04
Record Dates: First submitted 2022-07-06; First posted 2022-08-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Cancer Pain
MeSH Terms: conditions — Neoplasms; Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
observational , Monocentric, study to assess antalgic effects of well-being treatment in cancer care.

DETAILED DESCRIPTION:
Contrary to supportive care, well-being care is imperfectly assessed. Well being care (WBC) consist on complementary programs, with no real consensus. Very few studies have rigorously evaluated its benefits

The objective of this study was to evaluate the impact of four well-being treatments (foot reflexology, socio-aesthetics, Sophrology and singing) provided in a healthcare facility

ELIGIBILITY:
Inclusion Criteria:

* all type of cancer treated at the general Hospital of Valence
* patient agree to participate on Well being session: foot reflexology, socio-aesthetics, Sophrology and singing
* Age ≥ 18 years
* Affiliation to a Social security system
* Patient who has given written consent signed before any specific procedure of the protocol

Exclusion Criteria:

* Patient under guardianship, deprived of liberty, safeguard of justice
* Patient presenting a serious psychiatric pathology that does not allow compliance with the completion of the scale (at the discretion of the investigator)
* Refusal to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated for a cancer in CH Valence, agree to participate on one of the 4 Well being treatments: foot reflexology, socio-aesthetics, sophrology and singing
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Pain assesment | 1 immediately before well being treatment
  numerical scale 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."
Pain assesment | 1 immediately after well being treatment
  numerical scale 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Valence, Valence, Drome, France

IPD SHARING:
Plan to Share IPD: Undecided